CLINICAL TRIAL: NCT04579354
Title: Virtual Reality (VR) Tour to Reduce Preoperative Anxiety Before Anaesthesia in an Operating Setting: A Randomized Clinical Trial
Brief Title: Virtual Reality (VR) Tour to Reduce Preoperative Anxiety Before Anaesthesia
Acronym: VR OP- tour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EK037/20; CTC-A 20-026 (Other: RWTH Aachen)
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Anaesthesia; Anxiety; Postoperative Pain
Keywords: virtual reality (VR); anxiety preoperative; opearting theater
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Anaesthesia briefing (No Intervention): standardised anaesthesia information sessions, consisting of a detailed explanation of the anaesthesia procedure by the anaesthetist A specific information sheet is used to explain the procedure and the form of anaesthesia. This corresponds to the current procedure before an operation.
- Virtual reality (VR) tour (Experimental): standardised anaesthesia information sessions, consisting of a detailed explanation of the anaesthesia procedure by the anaesthetist A specific information sheet is used to explain the procedure and the form of anaesthesia.Subsequently, the patients are shown a virtual tour of the operation using VR glasses. This includes the way through the clinic to the operating theatre: Admission -> inpatient preparation for the operation -> administration of premedication -> way to the operating theater -> OP preparation (holding) -> safe surgery
  Interventions: Other: virtual reality tour

INTERVENTIONS:
Other: virtual reality tour — Patients will be guided via VR on their way through the hospital to the operating theater
  Arms: Virtual reality (VR) tour

SUMMARY:
Anxiety and apprehension are common among patients prior to surgery. This anxiety can lead to additional discomfort, increased pain sensation and increased stress symptoms. Virtual exposure has proven to be successful in exposure therapy for the treatment of the narrowest patients. Patients are not confronted with the real stimuli or situations that trigger the branches, but with virtual representations of them. Virtual reality (VR) makes it possible to create scenarios that would not be possible in reality because of the organisational, time or financial expenditure involved.The effectiveness of virtual stimulus exposure is well documented, especially in the case of object or situation-related fears in the context of specific phobias. It is therefore obvious that virtual stimulus exposure could also be suitable for minimising operation-associated fears.The research project described is designed to investigate the effect of virtual stimulus exposure on perioperative anxiety. For this purpose, a virtual tour of the operating setting has been created, which enables patients to explore the surroundings in detail by means of VR glasses.

DETAILED DESCRIPTION:
Anxiety and apprehension are common among patients prior to surgery. This anxiety can lead to additional discomfort, increased pain sensation and increased stress symptoms. Virtual exposure has proven to be successful in exposure therapy for the treatment of the narrowest patients. Patients are not confronted with the real stimuli or situations that trigger the branches, but with virtual representations of them. Virtual reality (VR) makes it possible to create scenarios that would not be possible in reality because of the organisational, time or financial expenditure involved.The effectiveness of virtual stimulus exposure is well documented, especially in the case of object or situation-related fears in the context of specific phobias. It is therefore obvious that virtual stimulus exposure could also be suitable for minimising operation-associated fears.The research project described is designed to investigate the effect of virtual stimulus exposure on perioperative anxiety. For this purpose, a virtual tour of the operating setting has been created, which enables patients to explore the surroundings in detail by means of VR glasses.

ELIGIBILITY:
Inclusion Criteria:

* all patient undergoing anaesthesia without the following exclusion criteria

Exclusion Criteria:

* < 18 years
* cancer surgery
* pregnancy
* postoperative setting ICU
* neurosurgery
* Thorax surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
STOA State T1 | before anaesthesia
  Questinaire STOA State T1 before anaesthesia

SECONDARY OUTCOMES:
STOA State T2 | within 48 hours after anaesthesia
  Questionaire STOA State T2 after anaesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogt L, Klasen M, Rossaint R, Goeretz U, Ebus P, Sopka S. Virtual Reality Tour to Reduce Perioperative Anxiety in an Operating Setting Before Anesthesia: Randomized Clinical Trial. J Med Internet Res. 2021 Sep 1;23(9):e28018. doi: 10.2196/28018. PMID 34252034